CLINICAL TRIAL: NCT06324357
Title: Beamion BCGC-1: A Phase Ib Dose Escalation and Phase II Dose Optimization, Randomized, Open-label, Multicenter Trial of Oral Zongertinib (BI 1810631) Alone or in Combination With Other Agents for the Treatment of Patients With Advanced HER2+ Metastatic Breast Cancer (mBC), Metastatic Gastric, Gastroesophageal Junction, or Esophageal Adenocarcinoma (mGEAC), or Metastatic Colorectal Cancer (mCRC)
Brief Title: Beamion BCGC-1: A Study to Find a Suitable Dose of Zongertinib Used Alone and in Combination With Other Treatments to Test Whether it Helps People With Different Types of HER2+ Cancer That Has Spread
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1479-0012
Record Dates: First submitted 2024-03-15; First posted 2024-03-21 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Breast Cancer; Metastatic Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma; Esophageal Adenocarcinoma; Colorectal Cancer
MeSH Terms: conditions — Breast Neoplasms; Adenocarcinoma Of Esophagus; Colorectal Neoplasms | interventions — trastuzumab deruxtecan; Ado-Trastuzumab Emtansine; Trastuzumab; Capecitabine; zanidatamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (18):
- Phase Ib - Cohort A: zongertinib + Trastuzumab emtansine (Experimental): Dose escalation (Phase Ib)
  Interventions: Drug: Zongertinib; Drug: Trastuzumab emtansine
- Phase Ib - Cohort B: zongertinib + Trastuzumab deruxtecan (Experimental): Dose escalation (Phase Ib)
  Interventions: Drug: Zongertinib; Drug: Trastuzumab deruxtecan
- Phase Ib - Cohort C: zongertinib + Trastuzumab deruxtecan (Experimental): Dose escalation (Phase Ib)
  Interventions: Drug: Zongertinib; Drug: Trastuzumab deruxtecan
- Phase II - Cohort D: zongertinib + Trastuzumab emtansine (Experimental): Dose optimization (Phase II).
  Interventions: Drug: Zongertinib; Drug: Trastuzumab emtansine
- Phase II - Cohort E: zongertinib + Trastuzumab deruxtecan (Experimental): Dose optimization (Phase II).
  Interventions: Drug: Zongertinib; Drug: Trastuzumab deruxtecan
- Phase II - Cohort F: zongertinib + Trastuzumab deruxtecan (Experimental): Dose optimization (Phase II).
  Interventions: Drug: Zongertinib; Drug: Trastuzumab deruxtecan
- Phase Ib - Cohort G: zongertinib + trastuzumab + capecitabine (Experimental): Dose escalation (Phase Ib)
  Interventions: Drug: Zongertinib; Drug: Trastuzumab; Drug: Capecitabine
- Phase Ib - Cohort K: zongertinib + trastuzumab (Experimental): Dose escalation (Phase Ib)
  Interventions: Drug: Zongertinib; Drug: Trastuzumab
- Phase II - Cohort H: zongertinib + trastuzumab + capecitabine (Experimental): Dose optimization (Phase II).
  Interventions: Drug: Zongertinib; Drug: Trastuzumab; Drug: Capecitabine
- Phase II - Cohort I: zongertinib (Experimental): Dose optimization (Phase II).
  Interventions: Drug: Zongertinib
- Phase II - Cohort J: zongertinib + trastuzumab (Experimental): Dose optimization (Phase II).
  Interventions: Drug: Zongertinib; Drug: Trastuzumab
- Phase II - Cohort I-ext: zongertinib (Experimental): Extension Phase II
  Interventions: Drug: Zongertinib
- Phase II - Cohort J-ext: zongertinib + trastuzumab (Experimental): Extension Phase II
  Interventions: Drug: Zongertinib; Drug: Trastuzumab
- Phase Ib - Cohort M: zongertinib + mFOLFOX6 (Experimental): Dose escalation (Phase Ib)
  Interventions: Drug: Zongertinib; Drug: mFOLFOX6
- Phase Ib - Cohort N: zongertinib + trastuzumab + mFOLFOX6 (Experimental): Dose escalation (Phase Ib)
  Interventions: Drug: Zongertinib; Drug: Trastuzumab; Drug: mFOLFOX6
- Phase Ib - Cohort O: zongertinib + zanidatamab (Experimental): Dose escalation (Phase Ib) - is not conducted in China or South Korea
  Interventions: Drug: Zongertinib; Drug: zanidatamab
- Phase II - Cohort L: zongertinib + trastuzumab (Experimental): Dose justification (Phase II)
  Interventions: Drug: Zongertinib; Drug: Trastuzumab
- Phase II - Cohort L-ext: zongertinib + trastuzumab (Experimental): Extension Phase II
  Interventions: Drug: Zongertinib; Drug: Trastuzumab

INTERVENTIONS:
Drug: Zongertinib — Zongertinib
  Other Names: BI 1810631, Hernexeos®
Drug: Trastuzumab deruxtecan — Trastuzumab deruxtecan
  Other Names: T-DXd; Enhertu®
  Arms: Phase II - Cohort E: zongertinib + Trastuzumab deruxtecan; Phase II - Cohort F: zongertinib + Trastuzumab deruxtecan; Phase Ib - Cohort B: zongertinib + Trastuzumab deruxtecan; Phase Ib - Cohort C: zongertinib + Trastuzumab deruxtecan
Drug: Trastuzumab emtansine — Trastuzumab emtansine
  Other Names: T-DM1; Kadcyla®
  Arms: Phase II - Cohort D: zongertinib + Trastuzumab emtansine; Phase Ib - Cohort A: zongertinib + Trastuzumab emtansine
Drug: Trastuzumab — Herceptin®
  Arms: Phase II - Cohort H: zongertinib + trastuzumab + capecitabine; Phase II - Cohort J-ext: zongertinib + trastuzumab; Phase II - Cohort J: zongertinib + trastuzumab; Phase II - Cohort L-ext: zongertinib + trastuzumab; Phase II - Cohort L: zongertinib + trastuzumab; Phase Ib - Cohort G: zongertinib + trastuzumab + capecitabine; Phase Ib - Cohort K: zongertinib + trastuzumab; Phase Ib - Cohort N: zongertinib + trastuzumab + mFOLFOX6
Drug: Capecitabine — Xeloda®
  Arms: Phase II - Cohort H: zongertinib + trastuzumab + capecitabine; Phase Ib - Cohort G: zongertinib + trastuzumab + capecitabine
Drug: mFOLFOX6 — mFOLFOX6
  Arms: Phase Ib - Cohort M: zongertinib + mFOLFOX6; Phase Ib - Cohort N: zongertinib + trastuzumab + mFOLFOX6
Drug: zanidatamab — zanidatamab
  Arms: Phase Ib - Cohort O: zongertinib + zanidatamab

SUMMARY:
This study is open to adults aged 18 years and older with different types of HER2+ cancer that has spread and cannot be removed by surgery. People can take part in this study if their tumours show HER2 aberrations and previous treatment was not successful. The purpose of this study is to find a suitable dose of zongertinib that people with different types of HER2+ cancer that has spread can tolerate best when taken together with trastuzumab deruxtecan (T-DXd), with trastuzumab emtansine (T-DM1), with trastuzumab and capecitabine, with zanidatamab, or with mFOLFOX6 (with or without trastuzumab). Another purpose is to check whether zongertinib alone and in combination with other treatments can make tumours shrink. Zongertinib inhibits HER2. HER2 causes cancer cells to grow.

In this study, participants receive treatment in cycles. Study participants are treated with zongertinib alone or in combination with other treatments. This study has 2 parts. In Part 1, participants in different groups receive increasing doses of zongertinib. In Part 2, participants are put into different groups by chance. Each group receives a different dose of zongertinib. Every participant has an equal chance of being in each group.

During the study, the participants visit the study site regularly. In this study, researchers want to find the highest dose of zongertinib that participants can tolerate when taken together with other treatments. To find this out, researchers look at certain severe health problems that a number of participants have. The doctors regularly check the size of the tumour with imaging methods (CT/MRI) during the study. The doctors also regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion criteria:

* Patients ≥18 years of age or over the legal age of consent in countries where that is greater than 18 years at the time of signature of the informed consent form (ICF)
* Cohorts A to K and Cohort O: Documented Human epidermal growth factor receptor 2 overexpressing and/or amplified (HER2+), metastatic breast cancer (mBC) or metastatic gastric adenocarcinoma, gastroesophageal junction adenocarcinoma, or esophageal adenocarcinoma (mGEAC).
* Cohorts L (L-ext), M, and N (metastatic colorectal cancer (mCRC)): Documented Human epidermal growth factor receptor 2 (HER2) overexpression/amplification according to American Society of Clinical Oncology/College of American Pathologists (ASCO/CAP) gastric cancer guidelines and according to the result of local testing.
* For dose optimization and justification (Phase II): Patient must provide tumor tissue from locations not radiated prior to biopsy, if possible, collected through archival tissue
* History of prior treatment lines in palliative setting:

  * For cohorts A, B, C, D, E, F, G, H, I, I-ext, J, J-ext, K and O documented investigator assessed progression after HER2-directed treatment for unresectable locally advanced or metastatic disease (For Cohorts D, H, I (I-ext), J (J-ext) - patients must have been pretreated with trastuzumab deruxtecan (T-DXd) and have progressed or have been intolerant to previous T-DXd).
  * For cohorts L, L-ext, M and N documented progression or recurrence of disease during or following their latest line of therapy. Patients must have had at least one prior line of therapy for locally advanced unresectable disease or metastatic disease (adjuvant and neoadjuvant therapy excluded) and documented disease progression or recurrence of disease during or following their latest line of therapy. In the opinion of the Investigator, patients must be unlikely to tolerate or derive clinically meaningful benefit from further standard of care therapy known to prolong survival.
* Presence of at least one measurable lesion according to RECIST 1.1
* Eastern Cooperative Oncology Group (ECOG) score of 0 or 1
* Adequate organ function based on laboratory values Further inclusion criteria apply.

Exclusion criteria:

* Previous treatment with:

  * Any small molecule HER2 inhibitor in the palliative setting in Cohorts D, E, F, H, L, L-ext, M, and N. In Cohort D allowed in up to 15 patients in each dose level (DL).
  * T-DXd in Cohorts E and F. In Cohort E allowed in up to 15 patients in each DL.
  * trastuzumab emtansine (T-DM1) in the palliative setting in Cohort D and H. In Cohort H allowed in up to 15 patients in each DL.
  * Capecitabine in Cohort D and H. In Cohort D allowed in up to 15 patients in each DL
* Presence of uncontrolled and/or symptomatic brain metastases, or leptomeningeal disease
* Mean resting corrected QT interval (QT interval corrected for heart rate by Fridericia´s formula (QTcF)) >470 msec.
* Any factors that increase the risk of QT interval corrected for heart rate (QTc) prolongation or risk of arrhythmic events such as heart failure, hypokalemia, congenital long QT syndrome, personal or family history of long QT syndrome or unexplained sudden death under 40 years-of-age.
* Ejection fraction <50% or the lower limit of normal of the institutional standard within 28 days prior to randomization
* History of (non-infectious) interstitial lung disease (ILD)/pneumonitis that required steroids, current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 768 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2029-01-08 (Estimated); Study Completion 2029-01-08 (Estimated)

PRIMARY OUTCOMES:
Dose escalation (Phase Ib): Occurrence of dose-limiting toxicities (DLTs) in the maximum tolerated dose (MTD) evaluation period | up to 21 days
  The MTD evaluation period is defined as the first 21 days of the first treatment cycle for Cohorts A, B, C, G, K, and O. The MTD evaluation period is defined as the first 28 days after the first administration of any trial medication for Cohorts M and N.
Dose optimization and justification (Phase II): Objective response (OR) | up to 50 months
  Objective response (OR) is defined as the best overall response of confirmed complete response (CR) or confirmed partial response (PR) according to RECIST 1.1 from the date of treatment start until the earliest date of disease progression, death, or last evaluable tumor assessment before start of subsequent anti-cancer therapy, or treatment discontinuation as assessed by investigator review.

SECONDARY OUTCOMES:
Dose escalation (Phase Ib): Objective response (OR) | up to 50 months
Dose escalation (Phase Ib): Occurrence of dose-limiting toxicities (DLTs) during the entire treatment period | up to 50 months
Dose escalation (Phase Ib): Maximum measured concentration of zongertinib (at steady state) (Cmax,(ss)) | up to 2 days
  For cycle 2 only.
Dose escalation (Phase Ib): Area under the concentration-time curve of zongertinib over the time interval from 0 to 4h at steady state (AUC0-4h,ss) | up to 2 days
  For cycle 2 only.
Dose escalation (Phase Ib): Area under the concentration-time curve of zongertinib over the time interval from 0 to the last quantifiable data point at steady state (AUC0-tz,ss) | up to 2 days
  For cycle 2 only.
Dose optimization and justification (Phase II): Progression-free survival (PFS) | up to 50 months
  PFS is defined as the time from treatment start until the earliest date of tumor progression according RECIST 1.1 based on investigator review or death from any cause, whichever occurs first.
Dose optimization and justification (Phase II): Disease control (DC) | up to 50 months
  DC is defined as best overall response of complete response (CR) or partial response (PR) or stable disease (SD) where best overall response is defined according to RECIST 1.1 from first treatment administration until the earliest of disease progression, death, or last evaluable tumor assessment before start of subsequent anti-cancer therapy, or treatment discontinuation, as assessed by investigator review.
Dose optimization and justification (Phase II): Occurrence of treatment-emergent AEs leading to zongertinib (BI 1810631) dose reduction during the on-treatment period | up to 50 months
Dose optimization and justification (Phase II): Maximum measured concentration (at steady state) (Cmax,(ss)) | up to 50 months
Dose optimization and justification (Phase II): Area under the concentration-time curve over the time interval from 0 to the last quantifiable data point at steady state (AUC0-tz,ss) | up to 50 months
Dose optimization and justification (Phase II): Patient-reported outcome (PRO) - PRO-CTCAE | up to 24 weeks
  The Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) item library was developed to elicit symptomatic toxicity information directly from patients in cancer clinical trials. The items selected for this trial are: Mouth/throat sores, Taste changes, Decreased appetite, Nausea, Vomiting, Constipation, Diarrhoea, Shortness of breath, Cough, Rash, Skin dryness, Hair loss, Itching, Numbness & Tingling, Fatigue, Nosebleed, Headache.
  PRO-CTCAE responses are scored from 0 (=none) to 4 (=very severe) (or 0/1 for absent/present).
Dose optimization and justification (Phase II): Patient-reported outcome (PRO) - EORTC IL46 | up to 48 weeks
  The EORTC IL46 is a single question that assesses bother (burden) of treatment. It is rated on a scale from 1 to 4, ranging from "not at all" to "very much".
Dose optimization and justification (Phase II): Patient-reported outcome (PRO) - EORTC IL19 | up to 48 weeks
  The EORTC IL19 consists of five physical functioning scale items. It is rated on a scale from 1 to 4, ranging from "not at all" to "very much".

CONTACTS AND LOCATIONS:
Locations (102):
- United States (25):
  - Mayo Clinic-Arizona, Phoenix, Arizona
  - The Oncology Institute of Hope and Innovation, Cerritos, California
  - Ellison Medical Institute, Los Angeles, California
  - Valkyrie Clinical Trials, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - University of California Irvine, Orange, California
  - Sharp Memorial Hospital, San Diego, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Mayo Clinic - Florida, Jacksonville, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Community Health Network, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Rochester, Minnesota
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Baptist Cancer Center - Memphis, Memphis, Tennessee
  - SCRI Oncology Partners, Nashville, Tennessee
  - Tennessee Oncology, Pllc, Nashville, Tennessee
  - The Methodist Hospital Research Institute, Houston, Texas
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Belgium (6):
  - Cliniques Universitaires Saint-Luc, Brussels
  - Edegem - UNIV UZ Antwerpen, Edegem
  - UZ Leuven, Leuven
  - Hôpital Vivalia De Libramont, Libramont-Chevigny
  - Centre Hospitalier Universitaire de Liège, Liège
  - CHU UCL Namur, Namur
- China (8):
  - Jilin Province Cancer Hospital, Changchun
  - The First Hospital of Jilin University, Changchun
  - Sir Run Run Shaw Hospital, Zhejiang University, School of Medicine, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Jiangsu Province Hospital, Nanjing
  - Fudan University Shanghai Cancer Center, Shanghai
  - Tianjin Cancer Hospital, Tianjin
  - Henan Cancer Hospital, Zhengzhou
- France (11):
  - INS Bergonie, Bordeaux
  - CTR François Baclesse, Caen
  - CTR Georges-François Leclerc, Dijon
  - CTR Leon Berard, Lyon
  - INS Paoli-Calmettes, Marseille
  - HOP Tenon, Paris
  - CTR Eugène Marquis, Rennes
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - Institut de Cancérologie de Strasbourg, Strasbourg
  - INS Claudius Regaud IUCT-Oncopole, Toulouse
  - INS Gustave Roussy, Villejuif
- Germany (6):
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Universitätsklinikum Erlangen, Erlangen
  - Evang. Kliniken Essen-Mitte gGmbh, Essen
  - Asklepios Kliniken GmbH & Co. KGaA, Hamburg
  - Universitätsklinikum Mannheim GmbH, Mannheim
  - Universitätsklinikum Ulm, Ulm
- Italy (8):
  - Istituto Di Candiolo, Candiolo (TO)
  - Az.Osp. Universitaria "Ospedali Riuniti", Foggia
  - Istituto Scientifico Romagnolo, Meldola (FC)
  - Ospedale San Raffaele S.r.l., Milan
  - Istituto Europeo di Oncologia, Milan
  - Humanitas Istituto Clinico Catanese S.p.A., Misterbianco (CT)
  - Istituto Nazionale IRCCS Tumori Fondazione Pascale, Napoli
  - Istituto Clinico Humanitas, Rozzano
- Japan (8):
  - Aichi Cancer Center Hospital, Aichi, Nagoya
  - Tokai University Hospital, Isehara
  - Hakuaikai Sagara Hospital, Kagoshima
  - Kanagawa Cancer Center, Kanagawa, Yokohama
  - National Cancer Center Hospital East, Kashiwa-shi
  - Kyoto University Hospital, Kyoto
  - Osaka International Cancer Institute, Osaka
  - Japanese Foundation for Cancer Research, Tokyo, Koto-ku
- South Korea (7):
  - CHA Bundang Medical Center, Seongnam-si
  - Seoul National University Bundang Hospital, Seongnam-si
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - The Catholic University of Korea, Seoul St.Mary's Hospital, Seoul
- Spain (14):
  - Hospital Teresa Herrera, A Coruña
  - Hospital del Mar, Barcelona
  - Hospital Universitari Vall D Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Duran i Reynals, L'Hospitalet de Llobregat
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Clínica Universidad de Navarra - Madrid, Madrid
  - Fundación Jiménez Díaz, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - CIO Clara Campal, Madrid
  - Hospital Universitario Virgen De La Macarena, Seville
  - Instituto Valenciano de Oncología, Valencia
- United Kingdom (9):
  - Velindre Cancer Centre, Cardiff
  - St James's University Hospital, Leeds
  - St Bartholomew's Hospital, London
  - University College Hospital, London
  - Royal Free Hospital, London
  - The Christie, Manchester
  - Freeman Hospital, Newcastle upon Tyne
  - Nottingham University Hospitals NHS Trust, Nottingham
  - The Royal Marsden Hospital, Sutton, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Hurvitz S, Simonelli M, Yarza R, Berz D, Kitano S, Del Conte G, Acosta Eyzaguirre D, Doger de Speville Uribe BG, Maier D, Erzen D, Aykut Yazgili S, Curigliano G, Deng T, Yan M, Zhang Q, Wang X, Nakayama I, Shitara K. Beamion BCGC-1: phase Ib/II trial of zongertinib for advanced HER2-positive breast or gastroesophageal cancers. Future Oncol. 2025 Nov;21(26):3385-3393. doi: 10.1080/14796694.2025.2569553. Epub 2025 Oct 17. PMID 41108088
- See also: Related Info — https://www.mystudywindow.com
- See also: Related Info — https://ascopubs.org/doi/10.1200/JCO.2025.43.4_suppl.TPS509
- See also: Related Info — https://www.esmoopen.com/article/S2059-7029(25)00849-X/fulltext#:~:text=Beamion%20BCGC-1%20%28NCT06324357%29%20is%20a%20Ph%20Ib%2FII%20trial,to%20ASCO-CAP%20guidelines%29%2C%20pretreated%20mBC%20will%20be%20enrolled.